CLINICAL TRIAL: NCT02115581
Title: Effect of Coenzyme Q10 (Ubiquinone) Supplementation on Ventricular Function of Children With Idiopathic Dilated Cardiomyopathy.A Randomised Clinical Trial
Brief Title: Coenzyme Q10 Supplementation in Children With Idiopathic Dilated Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tehran (Other)
Responsible Party: Principal Investigator, Giv Heidari-Bateni, Research Fellow, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CoenzymeQ10 and Cardiomyopathy
Record Dates: First submitted 2008-12-22; First posted 2014-04-16 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Dilated Cardiomyopathy
Keywords: Coenzyme O10; Children; Idiopathic Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coenzyme Q10 (Experimental): Known cases of idiopathic dilated cardiomyopathy who received supplementation of coenzyme Q10 as a part of their medical regimen.
  Dosage administered: 2 milligram/kilogram/day in 2 or 3 divided doses, these being increased to the maximum dose of 10 milligram/kilogram/day according to tolerance or the appearance of sideeffects.
  Interventions: Drug: Coenzyme Q10
- Placebo (Placebo Comparator): known cases of idiopathic dilated cardiomyopathy who received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coenzyme Q10 — dose of 2 mg/kg/day in 2 or 3 divided doses and increased to the maximum dose of 10 mg/kg/day according to the patient's tolerance
  Other Names: Ubiquinone
  Arms: Coenzyme Q10
Drug: Placebo — dose of 2 mg/kg/day in 2 or 3 divided doses and increased to the maximum dose of 10 mg/kg/day according to the patient's tolerance
  Other Names: no brand name
  Arms: Placebo

SUMMARY:
This study aims to determine the effect of Coenzyme Q10 supplementation on conventional therapy of children with heart failure due to idiopathic dilated cardiomyopathy.

DETAILED DESCRIPTION:
This study aims to determine the effect of Coenzyme Q10 supplementation on conventional therapy of children with heart failure due to idiopathic dilated cardiomyopathy. In a prospective, randomized, double-blinded, placebo-controlled trial, patients younger than 18 years with idiopathic dilated cardiomyopathy randomizes to receive either Coenzyme Q10 or placebo. Echocardiographic systolic and diastolic function parameters are determined for every patient at baseline, after three,six and nine months of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Known cases of Idiopathic Dilated Cardiomyopathy (IDC)
* Those patients in whom heart failure medications were stable for at least 1 month
* More than 6 months aged

Exclusion Criteria:

* Recent modification in medications
* Hemodynamic instability
* Congenital heart disease
* Metabolic heart disease
* Cardiac dysfunction resulting from abnormalities in other organs and those with an acquired cardiomyopathy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reza Shabanian, MD, Study Director — Children's Medical Center; Armen Kocharian, MD, Study Chair — Children's Medical Center; Giv Heidari-Bateni, MD/MPH, Principal Investigator — Children's Medical Center
Locations (1):
- Children's Medical Center, Tehran, Tehran Province, Iran

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients younger than 18 years with known diagnosis of primary dilated cardiomyopathy referred for follow-up echocardiography to Children's Medical Center between September 2006 to March 2008 were recruited.
Groups:
- Coenzyme Q10: Known cases of idiopathic dilated cardiomyopathy who received Co Q10
- Placebo: Known cases of idiopathic dilated cardiomyopathy who received the placebo
Period: Overall Study
Arm/Group | Coenzyme Q10 | Placebo
Started | 17 | 21
Completed | 17 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Conezyme Q10: known cases of idiopathic dilated cardiomyopathy who received Co Q10
- Total: Total of all reporting groups
Arm/Group | Conezyme Q10 | Placebo | Total
Number analyzed (Participants) | 17 | 21 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (4.5) | 7.3 (5.2) | 6.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 11 | 19
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 17 | 21 | 38

OUTCOME MEASURES:

1. Secondary Outcome: Adverse Events
Description: Number of patients with evidence of adverse reaction to coenzyme Q10 including nausea, vomiting, changes in blood pressure, neurological signs or any abnormal behavior like disquiet in young children.
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Conezyme Q10 | Placebo
Number analyzed (Participants) | 17 | 21
Participants | 0 | 0

2. Primary Outcome: Improvement in Left Ventricular Ejection Fraction
Description: Ejection Fraction of left ventricle (percentage of blood pumped out of left ventricle with each heart beat) calculated by echocardiography
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Conezyme Q10 | Placebo
Number analyzed (Participants) | 17 | 21
Percentage | 42.1 (14.7) | 37.6 (9.7)
Statistical Analysis 1: Comparison: Conezyme Q10 vs Placebo; Test type: Superiority or Other; p = 0.267, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Improvement in Left Ventricular Filling Abnormality
Description: Doppler-derived transmitral blood flow and pulmonary venous blood flow data were used for grading of the severity of diastolic filling abnormality in patients before and after the intervention. Diastolic filling abnormality was categorized as: 1- normal 2- abnormal relaxation 3- pseudonormal 4- restricted pattern based on echo data. The proportion of patients who showed improvement in the diastolic function grading was compared between the study groups.
Time Frame: 6 months
Measure: Number; unit: Percentage
Arm/Group | Conezyme Q10 | Placebo
Number analyzed (Participants) | 17 | 21
Percentage | 59 | 19
Statistical Analysis 1: Comparison: Conezyme Q10 vs Placebo; Test type: Superiority or Other; p = 0.011, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Coenzyme Q10 (Study Group): Known cases of idiopathic dilated cardiomyopathy
  Coenzyme Q10: dose of 2 mg/kg/day in 2 or 3 divided doses and increased to the maximum dose of 10 mg/kg/day according to the patient's tolerance
- Placebo (Control Group): Known cases of idiopathic dilated cardiomyopathy
  Placebo: dose of 2 mg/kg/day in 2 or 3 divided doses and increased to the maximum dose of 10 mg/kg/day according to the patient's tolerance
Arm/Group | Coenzyme Q10 (Study Group) | Placebo (Control Group)
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/21
Other Adverse Events (participants affected / at risk) | 0/17 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No